CLINICAL TRIAL: NCT04963491
Title: A Prospective Cohort Clinical Trial Study of Prosthesis and Surgery Guide System for Personalized Total Knee Arthroplasty
Brief Title: Prosthesis and Surgery Guide System for Personalized Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Inner Mongolia People's Hospital (Other); Jining Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2020518
Record Dates: First submitted 2021-06-17; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed personalized TKA prosthesis (Experimental): Design：Personalized TKA prosthesis Manufacture：3D
  Interventions: Device: Personalized TKA prosthesis
- Zimmer NexGen TKA prostheses (Active Comparator): Prosthesis has been widely used in clinic
  Interventions: Device: Zimmer NexGen prostheses

INTERVENTIONS:
Device: Personalized TKA prosthesis — TKA prosthesis that is designed and manufactured according to the patient's knee joint anatomy
  Arms: 3D printed personalized TKA prosthesis
Device: Zimmer NexGen prostheses — Commercial products used on a large scale
  Arms: Zimmer NexGen TKA prostheses

SUMMARY:
The subject is planned to carry out the clinical trails of femoral condyle prosthesis, tibial tray prosthesis and meniscus prosthesis; At the same time, in order to achieve personalized precision bone resection, the clinical trial verification is carried out on the personalized cutting guides.

DETAILED DESCRIPTION:
The subject continues the research of Professor Jia-kuo Yu's research group on the personalized design, processing and manufacturing of personalized total knee arthroplasty (TKA) prostheses and the verification of animal and human cadavers. It is planned to carry out the clinical trails of femoral condyle prosthesis, tibial tray prosthesis and meniscus prosthesis; At the same time, in order to achieve personalized precision bone resection, the clinical trial verification is carried out on the personalized cutting guides.

In the clinical validation study, the research team will summarize the role of personalized TKA prostheses and personalized TKA cutting guides in the precise and minimally invasive treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Degenerative osteoarthritis, traumatic arthritis or avascular necrosis, inflammatory joint disease and other end-stage knee joint diseases, as well as the correction of deformities, reconstruction after failure of some knee joint prostheses, and other techniques that cannot be handled In the case of fractures, total knee prosthesis replacement is required.
2. Age ≥50, ≤80 years old.
3. The subject or guardian is willing and able to sign an informed consent form.

Exclusion Criteria:

1. History of previous knee surgery.
2. Severe knee joint deformity (valgus greater than 15° or valgus greater than 20°) or knee joint instability;
3. Severe flexion contracture deformity (flexion contracture> 25°);
4. Perform total knee joint revision and replacement surgery;
5. Rheumatoid arthritis;
6. Body Mass Index (BMI) > 35.
7. Patients with neuromuscular insufficiency (for example, paralysis, myolysis or muscle weakness) can lead to postoperative knee instability or abnormal gait;
8. Pregnant or lactating women;
9. Suffer from the underlying medical condition (including but not limited to metabolism, hematology, kidney, liver, lung, nerve, endocrine, heart, infection or gastrointestinal tract) that the researcher believes that the patient is at an unacceptable risk; Serious progressive or uncontrolled diseases that are not suitable for trials or put them at high risk, including any medical or psychiatric conditions that the investigator believes will prevent subjects from following the protocol or completing the study according to the protocol.
10. Being infected with human immunodeficiency virus (HIV), infectious hepatitis B or hepatitis C, or a corresponding medical history.
11. Suffer from a progressive infection or malignant disease, and be able to provide chest X-ray, computed tomography (CT scan) or MRI evidence within 12 weeks before screening, and be verified by a qualified physician.
12. Active systemic infections (except colds) or any other infections that will recur regularly during the previous two weeks.
13. There is a history of chronic or recurrent infectious diseases, or evidence of tuberculosis infection that was judged to be positive at the time of screening. Subjects who have obtained positive or uncertain results can participate in the study if they have undergone a comprehensive tuberculosis examination (according to local practice/guidelines) within 12 weeks before baseline and finally confirmed that there is no evidence of active tuberculosis. If the presence of latent tuberculosis is confirmed, treatment must be initiated and maintained in accordance with local or national guidelines before the baseline.
14. History of lymphoproliferative disease, or any known malignant tumor, or history of malignant tumor of any organ system in the past 5 years (Bowen's disease, basal cell carcinoma, or actinic keratosis after treatment and no evidence of recurrence in the past 12 weeks Except for diseases; except for excised cervical carcinoma in situ or non-invasive malignant colon polyps).
15. At the same time suffering from medical problems, including but not limited to the following:
16. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥95mmHg), congestive heart failure (New York Heart Association status classification III or IV).
17. Subjects with a serum creatinine level exceeding 2.0 mg/dl (176.8 μmol/L).
18. Total white blood cell (WBC) count at screening <2500/μL, or platelet <100000/μL or neutrophil <1500/μL or hemoglobin <8.5 g/dL.
19. In the six months before the baseline, there is a history of alcohol or drug abuse or evidence of ongoing abuse.
20. The patient is mentally incapable or unable to understand the requirements for participating in the research.

Ages: 51 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical axis of the lower limb and prosthesis position | 7 days postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 3months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 6 months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 12 months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.

SECONDARY OUTCOMES:
Osteotomy during TKA | during surgery
  The size of the osteotomy
Operation time | during surgery
  operation time
VAS score | 7 days postoperatively
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 3months postoperatively
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 6 months postoperatively
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 12 months postoperatively
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
KSS score | 7 days postoperatively
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 3months postoperatively
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 6 months postoperatively
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 12 months postoperatively
  knee society score, the scale is 0-200 and 0 is worse.
WOMAC score | 7 days postoperatively
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 3months postoperatively
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 6 months postoperatively
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 12 months postoperatively
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
SF-36 score | 7 days postoperatively
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 3months postoperatively
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 6 months postoperatively
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 12 months postoperatively
  short form 36 questionnaire, scale is 0-100 and 0 is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No